CLINICAL TRIAL: NCT04502290
Title: Synchronized Brain and Hand Stimulation to Improve Hand Function After Stroke
Brief Title: Synchronized Brain and Hand Stimulation After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amit Sethi (Other)
Responsible Party: Sponsor-Investigator, Amit Sethi, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19070157
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Upper Extremity Paresis
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Combined non-invasive brain and Functional Electrical Stimulation (Experimental): In this arm of the study participants will receive repeated non-invasive brain stimulation synchronously paired with FES
  Interventions: Device: Combined Non-invasive brain stimulation and functional electrical hand stimulation

INTERVENTIONS:
Device: Combined Non-invasive brain stimulation and functional electrical hand stimulation — Participants will receive synchronously combined non-invasive brain stimulation (delivered via electrical/magnetic stimulation) with functional electrical stimulation (delivered via DS7A or Neuromove) of the weak hand

SUMMARY:
Among the 795,000 individuals who sustain a stroke annually in the United States, 65% continue to experience moderate-to-severe impairments in one hand six months or more, which limits their ability to perform daily tasks. Currently there is dearth of understanding of the mechanisms of motor recovery after stroke. Understanding the mechanisms can potentially lead to the development of interventions to improve motor performance after stroke. The proposed study will examine how synchronously pairing brain and hand stimulation repeatedly affects the plasticity of the brain and motor performance after stroke. The knowledge gained from this study can be useful to develop interventions to improve hand movement after moderate-severe stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (either right or left handed) with unilateral hemiparesis after stroke;
2. Stroke onset of at least six months prior to the time of participation;
3. Ability to elicit motor evoked potential in the Extensor digitorum communis (EDC) muscle
4. Ability to grasp, as indicated by a score of at least 1 (out of 2) on the finger mass flexion and cylindrical grasp items of Upper Extremity Fugl-Meyer scale
5. age between 18-80 years

Exclusion Criteria:

1. Presence of severe aphasia , measured by cognitive and/or language impairments that preclude the ability to follow simple instructions;
2. Excessive spasticity of wrist and finger muscles, defined as a Modified Ashworth Score more than or equal to 3, which may limit the ability to open the hand/fingers;
3. Diagnosis of neurological disorders other than stroke, which may confound the results;
4. Has touch and proprioceptive sensory deficits determined via a score of 0 on the position sense section (section H) of the Fugl Meyer Upper Extremity assessment proprioception, which may limit the ability to report excessive amount of tingling due to hand stimulation
5. History of seizure or epilepsy as the effects of TMS are not tested in individuals with seizures or epilepsy;
6. Orthopaedic/musculoskeletal conditions (eg, arthritis) affecting the upper extremity, which may limit the ability to move the affected hand
7. Presence of metallic implants in the head or neck for TMS;
8. Currently or planning to become pregnant, as the effects of TMS are not tested not pregnant women;
9. Difficulty maintaining alertness or remaining still for MRI;
10. Ferromagnetic metallic implants, pacemakers, other implanted devices, or ventilators (for MRI);
11. Bodyweight > 300 lbs due to MRI scanner dimensions
12. Psychiatric diagnosis according to the criteria of the Diagnostic and Statistical Manual of Mental Disorder, Fifth Edition (DSM-V), or who are on psychotropic medication, which may confound the results
13. Cognitive impairments, defined as a score of < 23 on the Mini Mental Status Examination, which may limit the ability to follow the commands in the study
14. Excessive pain > equal to 5 on Visual Analog Scale in the more-affected upper extremity, which may limit the ability to participate in the study
15. History of schizophrenia, Bipolar disorder (type I or II) [Answer yes to questions 16 and items of the (hypo) maniac module of the The Mini International Neuropsychiatric Interview], current moderate, severe depression (Scores of >10 on Patient Health Questionnaire-9) and other neurological or medical conditions that could confound results.
16. Life expectancy less than the duration of the study
17. Hemispatial neglect, which may limit the ability to pay attention to the affected hand
18. Participating in concurrent therapy, which may confound the results
19. We will exclude children because although stroke may occur in children, the protocol is addressing stoke in adults and the devices are not approved for use in children

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Sethi, Principal Investigator — UPitt
Locations (1):
- Neuromotor Recovery and Rehabilitation Lab, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 10 participants from 2020-2024.
Period: Overall Study
Arm/Group | Combined Non-invasive Brain and Functional Electrical Stimulation
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Combined Non-invasive Brain and Functional Electrical Stimulation
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Upper Limb Fugl-Meyer Score [Mean (Standard Deviation); unit: score on a scale] — This scale measures the motor control of the weak upper extremity after stroke. The minimum score is 0 and the maximum score is 66, where higher scores are considered as better motor control.
  score on a scale | 25 (5)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Box and Block Test
Description: The Box and Block Test (BBT) measures unilateral gross manual dexterity and the ability to release objects. It is a quick, simple and inexpensive test. It can be used with a wide range of populations, including clients with stroke. The BBT is composed of a wooden box divided in two compartments by a partition and 150 blocks. The BBT administration consists of asking the participants to move, one by one, the maximum number of blocks from one compartment of a box to another of equal size, within 60 seconds. The box is oriented lengthwise and placed at the client's midline, with the compartment holding the blocks oriented towards the hand being tested. Participants first perform this test with their unaffected hand in order to practice and register baseline scores. Additionally, a 15-second trial period is permitted at the beginning of each side. Before the trial, after the standardized instructions are given to participants are advised that their fingertips must cross the partition when
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: percent change of number of blocks
Arm/Group | Combined Non-invasive Brain and Functional Electrical Stimulation
Number analyzed (Participants) | 10
percent change of number of blocks | 20 (5)
Statistical Analysis 1: Comparison: Combined Non-invasive Brain and Functional Electrical Stimulation; Paired t-test was used, where null hypothesis stated that the percent change in the number of blocks after intervention will be not statistically significant; Test type: Superiority; p = .04, t-test, 2 sided

2. Secondary Outcome: Percent Change in Motor Evoked Potential
Description: Surface EMG electrodes (Ag-AgCl) will be applied to the belly of the affected EDC muscle and a reference electrode will be placed at the clavicle. The motor evoked potential (MEP) data will be collected by stimulating the targets in the grid at 2000 Hz with Signal software (CED, Cambridge, UK). The raw values are measured in mili volts, but we report as a percent change compared to the pre-intervention or baseline.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: percent change of motor evoked potential
Arm/Group | Combined Non-invasive Brain and Functional Electrical Stimulation
Number analyzed (Participants) | 10
percent change of motor evoked potential | 40 (7)
Statistical Analysis 1: Comparison: Combined Non-invasive Brain and Functional Electrical Stimulation; Paired t-test was used, where null hypothesis stated that the percent change in the motor evoked potnetial after intervention will be not statistically significant; Test type: Superiority; p = .02, t-test, 2 sided

3. Secondary Outcome: Average Percent Change in Hand Force
Description: We will measure force production of the combined wrist and finger extensors (EDC) using two 34.09 kg load cells embedded in cushioned customized platforms. The height of the load cells can be altered to accommodate individual hand sizes. Participants will perform 5 trials of combined isometric wrist and finger extension movements against load cells for 10 seconds. The force data will be amplified by 5-20K and collected at 1000 Hz using Biopac amplifier and software (Biopac Systems Inc, Goleta, CA, USA). To allow for the deliberate increase to peak force as well as the tendency to drop off near the end of the 10-second interval, we will calculate the combined wrist and finger extension force output over the central 5 second segment. We will average the force across 5 trials. The raw values are measured in kilograms force, but we report as an average percent change compared to the pre-intervention or baseline.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: percent change of force
Arm/Group | Combined Non-invasive Brain and Functional Electrical Stimulation
Number analyzed (Participants) | 10
percent change of force | 10 (2)
Statistical Analysis 1: Comparison: Combined Non-invasive Brain and Functional Electrical Stimulation; Paired t-test was used, where null hypothesis stated that the percent change in the force after intervention will be not statistically significant; Test type: Superiority; p = .04, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From enrollment until the end of 6 weeks
Description: There were no serious adverse events or any other adverse events reported. There was no all-cause mortality reported.
Arm/Group | Combined Non-invasive Brain and Functional Electrical Stimulation
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT04502290/Prot_SAP_003.pdf